CLINICAL TRIAL: NCT03895177
Title: Usefulness of Low kVp High mAs Computed Tomography for the Evaluation of Pancreatic Cancer Resectability
Brief Title: Evaluation of Resectability of Pancreatic Cancer Using Low kVp CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-2019-0140
Record Dates: First submitted 2019-03-06; First posted 2019-03-29 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Diagnoses Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low kVp high mAs CT group (Experimental): doing pancreatic CT with 80 kVp tube current with more than 500 mA tube current for the evaluation of pancreatic cancer resectability
  Interventions: Diagnostic Test: contrast enhanced computed tomography

INTERVENTIONS:
Diagnostic Test: contrast enhanced computed tomography — pancreatic protocol CT with 80kVp tube voltage and more than 500mA tube current acquire late arterial phase and portal venous phase using volus tracking method

SUMMARY:
The aim of this study is to investigate usefulness of low kVp high mAs computed tomography in evaluation of pancreatic cancer resectability.

ELIGIBILITY:
Inclusion Criteria:

* 1. age between 20 year-old and 85 year-old 2. patient with pancreatic cancer detected on standard CT scan using 120 kVp that obtained within one month 3. consider surgical resection for pancreatic cancer treatment 4. patients who can undergo contrast enhanced CT scan

Exclusion Criteria:

* 1. history of severe adverse reaction to iodine contrast 2. less than 60 of estimated GFR

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
accuracy of low kVp CT to assess R0 resection of pancreatic cancer | 2 weeks after surgery
  Pancreastic cancer resectability

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (6):
- South Korea (6):
  - Korea National Cancer Center, Goyang-si, Kyung-gi Do
  - Hallym University Sacred Heart Hospital, Anyang
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan medical Center, Seoul
  - Korea University Guro Hospital, Seoul